CLINICAL TRIAL: NCT02019147
Title: BiHiVE 2 Study. The Investigation and Validation of Predictive Biomarkers in Hypoxic-ischaemic Encephalopathy.
Brief Title: BiHiVE2 Study. The Investigation and Validation of Predictive Biomarkers in Hypoxic-ischaemic Encephalopathy.
Acronym: BiHiVE2
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Dr. Deirdre Murray, Senior Lecturer, Consultant Paediatrician, University College Cork
Other Study IDs: DM0113UCC
Record Dates: First submitted 2013-11-06; First posted 2013-12-24 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Hypoxic Ischaemic Encephalopathy (HIE); Asphyxia
Keywords: HIE; Biomarker
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Umbilical cord blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Term Hypoxic Ischaemic Encephalopathy: Term Hypoxic Ischaemic Encephalopathy (HIE)
- Healthy Term Neonates: Controls

SUMMARY:
Despite recent advances in the care of mothers and newborn infants, many infants (approximately 20 per 1000 live births) continue to need resuscitation at birth. A proportion of these infants will have sustained significant injury through interruption of their blood and oxygen supply prior to delivery (perinatal asphyxia). In 2-3 babies per 1000 this will lead to brain swelling and the risk of long term brain injury called neonatal hypoxic-ischaemic encephalopathy (HIE). HIE remains a cause of neonatal death and long term disability. Early and accurate prediction of outcome would allow us to intervene during the window of the first 6 hours following birth, prior to secondary reperfusion and secondary brain injury. Estimating severity of injury can be difficult in newborn infants. Condition at birth does not predict neonatal, or longer term outcome. Biomarkers which could be measured at the time of birth and analysed at the bedside would offer these infants the best chance of timely and effective intervention. Through the BIHIVE study we have identified a number of predictive biomarkers in hypoxic-ischaemic encephalopathy. These markers are present in umbilical cord blood and have been identified through proteomic and metabolomic analysis of a stored biobank of samples from a recruited cohort of infants with perinatal asphyxia and hypoxic-ischaemic encephalopathy. We now wish to validate these biomarkers in an additional cohort, and will continue to explore new biomarkers in our stored biobank of umbilical cord samples. In addition we wish to assess our ability to predict neurodevelopmental and behavioural outcome in these infants. In this way we will determine the most robust biochemical and clinical markers for the prediction of early and medium term outcome in HIE. This study will establish the evidence base and validation of these biomarkers to the point where they can be developed into a bedside diagnostic algorithm which can be used in the labour ward to immediately identify those infants at risk of HIE in time to prevent secondary damage.

DETAILED DESCRIPTION:
Background and current knowledge in the area:

Perinatal asphyxia is one of the commonest causes of neonatal death and long term disability, occurring in 20 per 1000 live births. Of these, approximately 2-3 per 1000 will go on to develop hypoxic-ischaemic encephalopathy (HIE) (1). In Ireland and the UK HIE is the third commonest cause of neonatal mortality, accounting for 9% of all deaths, and 21% of term deaths, while globally it is estimated to cause over 1 million neonatal deaths each year. For the survivors there is significant secondary morbidity associated, including cerebral palsy (15%), severe cognitive delay (11%), seizure disorders (8%), sensori-neural deafness (7%), and visual loss (3%)(2).

HIE is an evolving process, which can be simplified into two insults. The initial insult is significant cerebral hypoxia and/or ischaemia which is followed by energy depletion, from anaerobic metabolism leading to the accumulation of lactate, and loss of cellular integrity. This sets in motion a cascade of events with the resultant formation of free radicals, proteases and caspases leading to cell damage and apoptosis, the secondary insult(3). The secondary energy failure has been shown to occur between 6-48 hours after the initial insult.

Until recently no therapeutic intervention which could reduce the associated morbidity or mortality existed. However the recent publications of several international trials, and their subsequent meta-analysis has shown that early induced hypothermia is beneficial in HIE, improving survival and reducing neurological disability (4-5). Induced hypothermia has now become a standard of care in moderate/severe HIE. However to be effective it must be commenced within 6 hours of delivery, before the secondary energy failure occurs. In this narrow window of time the population who would benefit from treatment must be identified, resuscitated, stabilised and cooled.

Unfortunately the ability to recognise and diagnose those who would benefit from therapy is not always possible within this time period. We have shown that the current standard methods to identify those at risk of HIE such as acid-base balance, lactate and Apgar score and initial neurological assessment are unreliable (6). Neonatal electroencephalography (EEG) is useful for the grading of encephalopathy and is an excellent predictor of long term outcome. In particular its evolution over the first 24 hours following delivery strongly correlates with outcome (7). However it requires a highly specialised skill set that is rarely available to the neonatologist in the acute setting. Amplitude integrated EEG is more widely used by clinicians, but its interpretation is user dependent, and the majority of neonatologists report they are not confident in their own interpretive ability (8). The need for early and reliable prediction of outcome in HIE has never been greater. A quick, cheap, reproducible, non-user dependent method for quantifying severity of HIE and likely prognosis is an urgent need. Many biochemical and haematological markers have been proposed in perinatal asphyxia, but none have led to clinical advances, or commercially viable bedside tests (9).

Over the last 2 years, here in the Cork University Maternity Hospital, through the BIHIVE study (Biomarkers in Hypoxic-Ischaemic Encephalopathy study) we have identified potential biochemical markers in umbilical cord blood which can accurately identify those infants who will progress to moderate/severe encephalopathy (10,11). The BIHIVE study has adopted a multifaceted approach to identifying blood-borne biomarkers in HIE through 1) targeted proteomic profiling using Luminex technology 2) miRNA profiling 3) comprehensive mapping of the blood metabolome using both Mass Spectrometry and Nuclear Magnetic Resonance techniques.

Our aim is to recruit a cohort of infants with clearly defined perinatal asphyxia and HIE, classified using both repeated neurological assessment and multichannel EEG. At the time of birth, umbilical cord blood will be drawn, processed and banked, using strict standard operating procedures (SOPs) which we have developed for this purpose. These procedures will ensure that all specimens will be suitable for later proteomic, metabolomic, transcriptomic and genomic analysis. Using a systems biology approach we have studied multiple proposed markers in the stored umbilical cord blood from our discovery cohort, initially focusing on the proteome and metabolome. Through this work we have already identified a number of biomarkers present in umbilical cord blood with the potential to predict the development of moderate/severe HIE. Our early data is extremely promising. Our initial metabolomic analysis has shown that we can differentiate between HIE and controls with an area under the curve (AUROC) of 0.92. Further analysis will be required to identify and quantify the exact metabolite peaks which produce this differentiation. We now wish to validate these findings in a further cohort of infants with perinatal asphyxia and HIE, and to validate our ability to predict longer term neurological outcome. Our pilot work examining microRNA changes in the cord blood of infants with moderate/severe HIE is also very encouraging with significant upregulation of a multiple studied miRNAs in both asphyxia and HIE. The most promising miRNAs are now being quantified using polymerase chain reaction (PCR) amplication and will be validated in the discovery cohort.

Future cohort-BIHIVE2: To develop these markers further to the point where we have validated a marker with >90% sensitivity and specificity for moderate/severe HIE we will need to recruit a further cohort of carefully recruited infants with high quality biobanking at birth and detailed clinical phenotyping. This is the main work of this current application. We will require a further cohort of 300 infants with perinatal asphyxia, of whom 60 will develop HIE and 30 will develop moderate to severe HIE. We will also need to recruit 300 contemporary control infants. To recruit this number of infants with perinatal asphyxia we will need to study 30,000 live births. We have therefore expanded our study centres to include Karolinska University Hospital, Stockholm, a large state of the art maternity hospital with 10,000 live births per annum.

Further validation will allow us to develop an algorithm of clinical and biochemical markers which will provide a sensitive and specific predictive test for moderate/severe HIE. Neurodevelopmental follow up of both cohorts will allow us to assess our ability to predict neurodevelopmental and behavioural outcome at 2 years.

Lastly we will examine the exact timing of biomarker alteration using a timed animal model of hypoxic-ischaemic injury (HI). In clinical studies hypoxic-ischaemic injury is unpredictable and its timing is often impossible to estimate. Dr Tracey Bjorkmann in Queen's University, Brisbane has developed a piglet model of HI which produces HI induces seizures and a level of injury equating to moderate to severe HIE (12). She has agreed to collaborate with our programme and will provide piglet samples of serum taken at 0,1,2 and 12 hours following HI. These samples will be invaluable in examining the progression of biomarker derangement and will help us to time neonatal brain injury after delivery.

ELIGIBILITY:
Inclusion Criteria:

Term infants defined at greater than 36 weeks gestation

All infants with one or more of the following clinical markers of HIE:

Apgar score less than or equal to 6 at 5 minutes pH < 7.1 on cord blood, Requiring intubation or CPR at birth -

Exclusion Criteria:

Outborn babies Less than 36 weeks gestation

-

Max Age: 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term Neonates born in hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
EEG confirmed hypoxic-ischaemic brain injury in the first 72 hours of life | 24 hours
  Clinical examination using the Thompson Encephalopathy score and visual interpretation of multichannel EEG

SECONDARY OUTCOMES:
Neurodevelopmental outcome at 2 years of age assessed using BSID III | 18-24 months
  Bayley's Scales of infant Development Version III

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Murray, MD, Principal Investigator — University College Cork, Ireland
Locations (2):
- Cork University Maternity Hospital, Cork, Ireland
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Conway JM, Walsh BH, Boylan GB, Murray DM. Mild hypoxic ischaemic encephalopathy and long term neurodevelopmental outcome - A systematic review. Early Hum Dev. 2018 May;120:80-87. doi: 10.1016/j.earlhumdev.2018.02.007. Epub 2018 Feb 26. PMID 29496329
- [Background] O'Connor CM, Ryan CA, Boylan GB, Murray DM. The ability of early serial developmental assessment to predict outcome at 5years following neonatal hypoxic-ischaemic encephalopathy. Early Hum Dev. 2017 Jul;110:1-8. doi: 10.1016/j.earlhumdev.2017.04.006. Epub 2017 Apr 21. PMID 28433953
- [Background] Murray DM, O'Connor CM, Ryan CA, Korotchikova I, Boylan GB. Early EEG Grade and Outcome at 5 Years After Mild Neonatal Hypoxic Ischemic Encephalopathy. Pediatrics. 2016 Oct;138(4):e20160659. doi: 10.1542/peds.2016-0659. Epub 2016 Sep 20. PMID 27650049
- [Background] Denihan NM, Boylan GB, Murray DM. Metabolomic profiling in perinatal asphyxia: a promising new field. Biomed Res Int. 2015;2015:254076. doi: 10.1155/2015/254076. Epub 2015 Jan 31. PMID 25802843
- [Background] Ahearne CE, Boylan GB, Murray DM. Short and long term prognosis in perinatal asphyxia: An update. World J Clin Pediatr. 2016 Feb 8;5(1):67-74. doi: 10.5409/wjcp.v5.i1.67. eCollection 2016 Feb 8. PMID 26862504
- [Result] Walsh BH, Broadhurst DI, Mandal R, Wishart DS, Boylan GB, Kenny LC, Murray DM. The metabolomic profile of umbilical cord blood in neonatal hypoxic ischaemic encephalopathy. PLoS One. 2012;7(12):e50520. doi: 10.1371/journal.pone.0050520. Epub 2012 Dec 5. PMID 23227182
- [Result] Walsh BH, Boylan GB, Dempsey EM, Murray DM. Association of nucleated red blood cells and severity of encephalopathy in normothermic and hypothermic infants. Acta Paediatr. 2013 Feb;102(2):e64-7. doi: 10.1111/apa.12086. Epub 2012 Dec 7. PMID 23157330
- [Result] Denihan NM, Kirwan JA, Walsh BH, Dunn WB, Broadhurst DI, Boylan GB, Murray DM. Untargeted metabolomic analysis and pathway discovery in perinatal asphyxia and hypoxic-ischaemic encephalopathy. J Cereb Blood Flow Metab. 2019 Jan;39(1):147-162. doi: 10.1177/0271678X17726502. Epub 2017 Aug 25. PMID 28840775
- [Result] Ahearne CE, Chang RY, Walsh BH, Boylan GB, Murray DM. Cord Blood IL-16 Is Associated with 3-Year Neurodevelopmental Outcomes in Perinatal Asphyxia and Hypoxic-Ischaemic Encephalopathy. Dev Neurosci. 2017;39(1-4):59-65. doi: 10.1159/000471508. Epub 2017 May 11. PMID 28490023
- [Result] Looney AM, Ahearne CE, Hallberg B, Boylan GB, Murray DM. Downstream mRNA Target Analysis in Neonatal Hypoxic-Ischaemic Encephalopathy Identifies Novel Marker of Severe Injury: a Proof of Concept Paper. Mol Neurobiol. 2017 Dec;54(10):8420-8428. doi: 10.1007/s12035-016-0330-4. Epub 2016 Dec 12. PMID 27957679
- [Result] Ahearne CE, Denihan NM, Walsh BH, Reinke SN, Kenny LC, Boylan GB, Broadhurst DI, Murray DM. Early Cord Metabolite Index and Outcome in Perinatal Asphyxia and Hypoxic-Ischaemic Encephalopathy. Neonatology. 2016;110(4):296-302. doi: 10.1159/000446556. Epub 2016 Aug 3. PMID 27486995
- [Result] Looney AM, Ahearne C, Boylan GB, Murray DM. Glial Fibrillary Acidic Protein Is Not an Early Marker of Injury in Perinatal Asphyxia and Hypoxic-Ischemic Encephalopathy. Front Neurol. 2015 Dec 21;6:264. doi: 10.3389/fneur.2015.00264. eCollection 2015. PMID 26733938
- [Result] Looney AM, Walsh BH, Moloney G, Grenham S, Fagan A, O'Keeffe GW, Clarke G, Cryan JF, Dinan TG, Boylan GB, Murray DM. Downregulation of Umbilical Cord Blood Levels of miR-374a in Neonatal Hypoxic Ischemic Encephalopathy. J Pediatr. 2015 Aug;167(2):269-73.e2. doi: 10.1016/j.jpeds.2015.04.060. Epub 2015 May 19. PMID 26001314
- [Result] Denihan NM, Walsh BH, Reinke SN, Sykes BD, Mandal R, Wishart DS, Broadhurst DI, Boylan GB, Murray DM. The effect of haemolysis on the metabolomic profile of umbilical cord blood. Clin Biochem. 2015 May;48(7-8):534-7. doi: 10.1016/j.clinbiochem.2015.02.004. Epub 2015 Feb 16. PMID 25697106
- [Result] Reinke SN, Walsh BH, Boylan GB, Sykes BD, Kenny LC, Murray DM, Broadhurst DI. 1H NMR derived metabolomic profile of neonatal asphyxia in umbilical cord serum: implications for hypoxic ischemic encephalopathy. J Proteome Res. 2013 Sep 6;12(9):4230-9. doi: 10.1021/pr400617m. Epub 2013 Aug 21. PMID 23931672
- [Result] Denihan NM, Looney A, Boylan GB, Walsh BH, Murray DM. Normative levels of Interleukin 16 in umbilical cord blood. Clin Biochem. 2013 Dec;46(18):1857-9. doi: 10.1016/j.clinbiochem.2013.07.012. Epub 2013 Jul 24. PMID 23891891
- [Result] Walsh BH, Boylan GB, Livingstone V, Kenny LC, Dempsey EM, Murray DM. Cord blood proteins and multichannel-electroencephalography in hypoxic-ischemic encephalopathy. Pediatr Crit Care Med. 2013 Jul;14(6):621-30. doi: 10.1097/PCC.0b013e318291793f. PMID 23823198